CLINICAL TRIAL: NCT02622958
Title: A Feasibility Study for a Phase 3, Randomized, Four-Week, Double-Blind, Placebo-Controlled, Crossover Trial of the Efficacy and Safety of PH94B Nasal Spray in the Acute Treatment of Social Anxiety Disorder (SAD)
Brief Title: Feasibility Study of PH94B Nasal Spray for Acute Treatment of Social Anxiety Disorder (SAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pherin Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PH94B CL028
Record Dates: First submitted 2014-03-18; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Social Phobia; Performance Anxiety; Social Anxiety; Anxiety
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PH94B Nasal Spray (Experimental): Water based solution of 16 ppm PH94B. Each nasal spray delivers .8 micrograms PH94B in 50 microliters
  Interventions: Drug: PH94B
- Placebo Nasal Spray (Placebo Comparator): Water based solution, each nasal spray delivers 50 microliters of droplets.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PH94B — PH94B is self-administered intranasally as needed or as necessary, no more than four doses per day for male and female subjects. Each spray delivers 50 µL (0.8 µg PH94B).
  Dosing is sex-specific:
  * Males: two (2) sprays (100 µL) are to be administered to each nostril, for a total dose of 3.2 µg
  * Females: one (1) spray (50 µL) is to be administered to each nostril, for a total dose of 1.6 µg
  Arms: PH94B Nasal Spray
Other: Placebo — Placebo is self-administered intranasally as needed or as necessary, no more than four doses per day for male and female subjects. Each spray delivers 50 µL (0.8 µg Placebo).
  Dosing is sex-specific:
  * Males: two (2) sprays (100 µL) are to be administered to each nostril, for a total dose of 3.2 µg
  * Females: one (1) spray (50 µL) is to be administered to each nostril, for a total dose of 1.6 µg
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of the study is to determine whether the PH94B nasal spray is effective for Acute Treatment of the symptoms of Social Anxiety Disorder (SAD) in adult men and women. The hypothesis is that PH94B nasal spray (.8 micrograms) has a rapid onset of efficacy to improve performance and interaction anxiety in patients with diagnosed Social Anxiety Disorder (SAD).

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled, 2-way crossover trial of the efficacy and safety of PH94B in the treatment of subjects diagnosed with Social Anxiety Disorder as defined by the Diagnostic and Statistical Manual IV and confirmed by the MINI (5.0.0). The study is intended to serve as a feasibility trial of a multi-center phase 3 study protocol of similar design.

The primary objective of this study is to evaluate design features for a larger Phase 3 study that will evaluate the safety and efficacy of PH94B for the acute management of symptoms in subjects with Social Anxiety Disorder. Careful review of diary entries and measurement of study medication compliance each week will be used to determine the feasibility of using the study medication on an "as needed" basis for anxiety-provoking social events. Specifically, the frequency of use, variability of SUDS ratings, effect size of differences in average peak SUDS ratings during treatment with PH94B and placebo, and general reliability of the diary recording method will be evaluated and used to refine inclusion and exclusion criteria as well as provide guidance for designing a larger multi-site study.

The study will last a total of 6-8 weeks. The randomized double-blind treatment period will last a total of four weeks for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to conducting any study-specific assessment.
* Male and female adults, 18 through 65 years of age, inclusive.
* Current diagnosis of Social Anxiety Disorder as defined in the DSM IV of Mental Disorders, which is not secondary to another pre-existing psychiatric condition or to a medical condition.
* Confirmation of diagnosis of Social Anxiety Disorder according to the MINI, 5.0.0
* Clinician-rated Liebowitz Social Anxiety Scale total score ≥60 at both Screening and Baseline visits.
* Clinician-rated HAM-D17 total score <18 at both Screening and Baseline visits.
* CGI-Severity score ≥4 at both Screening and Baseline visits.
* Subject must have:

  * experienced and documented a minimum total of six social interaction or performance events during the two week Screening Period prior to the Baseline Visit, and
  * for at least three of these events, must have achieved a peak score of ≥60 on the Subjective Units of Distress Scales (SUDS), as rated in the Patient Diary.
* Women of child-bearing potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the study and have a negative urine pregnancy test result prior to study medication administration.

Exclusion Criteria:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, eating disorder, obsessive-compulsive disorder. Any other current Axis I disorder other than SAD which is the primary focus of treatment. Note that subjects with concurrent Generalized Anxiety Disorder (GAD) are eligible for the study provided that GAD is not the primary diagnosis.
* Subjects who meet criteria for substance abuse within the year prior to entry.
* Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, or nasal-septal perforation that may have damaged the nasal chemosensory epithelium.
* An acute or chronic condition, including an infectious illness, uncontrolled seasonal allergies at the time of the study, or significant nasal congestion that potentially could affect drug delivery to the nasal chemosensory epithelium.
* Two or more documented failed treatment trials with a registered medication approved for SAD during the previous six months, whereby a treatment trial is defined as a period of at least six (6) weeks (or longer as documented in package insert for a particular drug) during which the patient received an adequate dosage (defined as the treatment dose indicated in the package insert to obtain efficacy for that particular drug) of the medication.
* Use of any psychotropic medication within 30 days prior to study entry (other than eszopiclone, ramelteon, zaleplon, or zolpidem for insomnia as described in Section 3.3).
* Concomitant use of non-study anxiolytics such as benzodiazepines or beta blockers during the study and within 30 days prior to study entry.
* Concomitant use of any over-the-counter, prescription product, or herbal preparation for treatment of the symptoms of social anxiety during the study and within 30 days prior to study entry.
* Prior exposure to PH94B.
* Improvement of more than 20% in the LSAS score at Baseline relative to Screening.
* Women who have a positive urine human chorionic gonadotropin pregnancy test prior to study medication administration.
* Subjects with clinically significant abnormalities in hematology, blood chemistry, urinalysis, ECG, or physical examination identified at the Screening or Baseline visit.
* Subjects with a positive urine drug screen at either the Screening or Baseline visit.
* Presence of any clinical condition or disease, or use of a concomitant medication, that in the clinical judgment of the Investigator could place the patient at undue risk, interfere with study participation, or confound the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subjective units of distress | Study medication nasal spray is to be administered 15 minutes prior to public performance and following each event they will be asked to record maximum subjective anxiety level experienced during the event.
  The primary study endpoint is average peak anxiety level for public performance or social interaction events during the two 2-week double-blind treatment phases (PH94B and placebo). Subjects will be asked to self-administer double-blind PH94B or placebo 15 minutes prior to public performance or social interaction events. Following each event, they will be asked to record the maximum (peak) subjective anxiety level experienced during the event using the patient rated Subjective Units of Distress Scale (SUDS), where anxiety scores range from 0 (no anxiety) to 100 (maximum anxiety ever experienced). Within each 2-week treatment phase, all subjective anxiety ratings will be summed and divided by the number of events recorded.

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement rating & Liebowitz Social Anxiety Scale | At baseline and following 2 weeks of treatment with Study medication nasal spray
  Two key secondary endpoints of the study are overall subject improvement as assessed by the Clinical Global Impression of Improvement rating (CGI-I), and the Investigator rated Liebowitz Social Anxiety Scale (LSAS). The proportion of subjects receiving a clinician-rated CGI-I score of 1 (Very much improved) or 2 (Much improved) following two weeks of treatment with placebo will be compared to the proportion of patients receiving a clinician-rated CGI-I score of 1 or 2 following two weeks of treatment with PH94B.

OTHER OUTCOMES:
Changes from screening/baseline in clinical laboratory values, ECGs, physical examinations, and vital sign assessments. | Every two weeks during treatment and one week after treatment with Study Medication Nasal Spray
  Safety and tolerability of PH94B will be assessed through changes from screening/baseline in laboratory values, ECGs, physical examinations, and vital sign assessments following exposure to PH94B, as well as by comparison of adverse events reported during treatment with PH94B and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Liebowitz, Principal Investigator — The Medical Research Network
Locations (1):
- The Medical Research Network, LLC, New York, New York, United States

REFERENCES:
- [Derived] Liebowitz MR, Hanover R, Draine A, Lemming R, Careri J, Monti L. Effect of as-needed use of intranasal PH94B on social and performance anxiety in individuals with social anxiety disorder. Depress Anxiety. 2016 Dec;33(12):1081-1089. doi: 10.1002/da.22546. Epub 2016 Aug 25. PMID 27561175